CLINICAL TRIAL: NCT00090051
Title: Open-label, Multicenter, Randomized, Comparative, Phase III Study to Evaluate the Efficacy and Safety of FCR vs. FC Alone in Previously Treated Patients With CD20 Positive B-cell CLL
Brief Title: FCR Versus FC Alone in the Treatment of Chronic Lymphocytic Leukemia (CLL) in Relapsed Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Biogen (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-14; BO17072
Record Dates: First submitted 2004-08-23; First posted 2004-08-25 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine+Cyclophosphamide (FC) (Active Comparator)
  Interventions: Drug: Fludarabine Phosphate; Drug: Cyclophosphamide
- Fludarabine+Cyclophosphamide+Rituximab (FCR) (Experimental)
  Interventions: Drug: Rituximab; Drug: Fludarabine Phosphate; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Rituximab — Intravenous repeating dose
  Arms: Fludarabine+Cyclophosphamide+Rituximab (FCR)
Drug: Fludarabine Phosphate — Intravenous repeating dose
Drug: Cyclophosphamide — Intravenous repeating dose

SUMMARY:
The purpose of this study is to provide treatment for patients who have chronic lymphocytic leukemia (CLL), and to compare the use of rituximab added to fludarabine+cyclophosphamide (FC) with FC alone, to determine if rituximab lengthens the time a patient remains free of leukemia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Established diagnosis of B-cell CLL by NCI Working Group criteria
* ≤1 previous line of chemotherapy
* Expected survival >6 months
* Acceptable hematologic status, liver function, renal function, and pulmonary function
* Negative serum pregnancy test for both pre-menopausal women and for women who are < 2 years after the onset of menopause
* Written informed consent

Exclusion Criteria:

* Prior treatment with interferon, rituximab or other monoclonal antibody
* Prior allogeneic bone marrow transplant (BMT) or autologous BMT or peripheral stem cell transplant (PBSCT) or patients who are considered to be candidates for allogeneic or autologous BMT or PSCT as assessed by their treating physician
* Fertile men or women of childbearing potential not using adequate contraception
* Severe Grade 3 or 4 non-hematological toxicity or prolonged (> 2 weeks) Grade 3 or 4 cytopenia on prior fludarabine or nucleoside analogue regimen
* History of fludarabine-induced or clinically significant autoimmune cytopenia
* History of other malignancies within 2 years prior to study entry, except for adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low-grade early stage localized prostate cancer treated surgically with curative intent; good prognosis ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone with curative intent.
* Medical conditions requiring long term use (> 1 month) of systemic corticosteroids
* Active bacterial, viral, or fungal infection requiring systemic therapy
* Severe cardiac disease
* Seizure disorders requiring anticonvulsant therapy
* Severe chronic obstructive pulmonary disease with hypoxemia
* Uncontrolled diabetes mellitus or hypertension
* Transformation to aggressive B-cell malignancy.
* Known infection with HIV, HCV, or hepatitis B
* Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to entering this study
* Known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
* Any co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2003-07-31 (Actual); Primary Completion 2008-07-23 (Actual); Study Completion 2012-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (106):
- United States (6):
  - Uab Comprehensive Cancer Center, Birmingham, Alabama
  - Pacific Coast Hematology/Oncology Medical Group, Fountain Valley, California
  - California Cancer Center Woodward Park; Community Medical Centers, Fresno, California
  - Rush-Presbyterian St. Luke'S Medical Center, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Milton S. Hershey Medical Center; Penn State Cancer Inst., Hershey, Pennsylvania
- Australia (4):
  - Concord Repatriation General Hospital; Haematology, Sydney, New South Wales
  - Mater Hospital; Division of Cancer Services, Brisbane, Queensland
  - Frankston Hospital; Oncology/Haematology, Frankston, Victoria
  - Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - Institut Jules Bordet, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Canada (9):
  - Uni of Alberta Hospital, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - QEII HSC; Oncology, Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Cancer Centre; Hematology, Hamilton, Ontario
  - The Ottawa Regional Hospital - General Campus; Division of Hematology, Box 704, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
- Denmark (2):
  - Aarhus Universitetshospital, Hæmatologisk Afdeling R, Aarhus
  - Righospitalet, Hæmatologisk Klinik, København Ø
- France (19):
  - Hopital Avicenne; Hematologie Biologique, Bobigny
  - Hopital Clemenceau; Hematologie Clinique, Caen
  - Chu Estaing; Hematologie Clinique Adultes, Clermont-Ferrand
  - Hopital Henri Mondor; Hematologie Clinique, Créteil
  - Clinique Victor Hugo; Chimiotherapie, Le Mans
  - Hopital Claude Huriez; Hematologie, Lille
  - Hopital Edouard Herriot; Bat.E-Hematologie, Lyon
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut J Paolii Calmettes; Onco Hematologie 1, Marseille
  - Hôpital Lapeyronie; Hématologie Oncologie Médicale, Montpellier
  - Hopital Hotel Dieu Et Hme;Hopital De Jour, Nantes
  - Hotel Dieu; Hematologie- Oncologie, Paris
  - Inserm Cic 9504, Paris
  - Hopital Pitie Salpetriere; Hematologie Clinique, Paris
  - Ch Lyon Sud; Hemato Secteur Jules Courmont, Pierre-Bénite
  - Chu La Miletrie; Hdj Cons Hemato Cancerologie, Poitiers
  - Centre Henri Becquerel; Hematologie, Rouen
  - Hopital Bretonneau; Clinique D'Oncologie & de Radiotherapie, Tours
  - Hopitaux De Brabois; Hematologie Medecine Interne, Vandœuvre-lès-Nancy
- Hungary (7):
  - Szent Laszlo Hospital; Hematology Dept, Budapest
  - National Institute of Oncology, A Dept of Internal Medicine, Budapest
  - Országos Gyógyintézeti Központ; Haematologiai Osztaly, Budapest
  - Uni of Debrecen; 2Nd Clinic of Internal Medicine, Debrecen
  - University of Debrecen Medical and Health Science Center, Institute of Internal Medicine, Hematology, Debrecen
  - Uni of Pecs; Dept of Internal Medicine, Pécs
  - University of Szeged, II Dept of Internal Medicine, Szeged
- Italy (10):
  - Uni Degli Studi Di Bari, Policlinico; Cattedra Di Ematologia,Dipart. Di Medicina Interna E Publica, Bari, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Ematologia E Trapianto Di Midollo Osseo, San Giovanni Rotondo, Apulia
  - A.O. Universitaria Federico II Di Napoli; Oncologia Ed Endocrinologia Clinica, Napoli, Campania
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - Ospedale S. Eugenio; Divisione Di Ematologia, Rome, Lazio
  - Az. Osp. S. Camillo Forlanini; Uo Ematologia E Trapianti Di Midollo Osseo, Rome, Lazio
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia;Dip. Biotecnologie Cel CELLULARI ED EMATOLOGIA, Rome, Lazio
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Ospedale Di Vicenza; Nefrologia, Ematologia, Vicenza, Veneto
- Netherlands (4):
  - Meander Mc, Locatie Lichtenberg; Dept of Lung Diseases, Amersfoort
  - Academisch Medisch Centrum Universiteit Amsterdam, Amsterdam
  - Erasmus Mc - Daniel Den Hoed Kliniek; Medical Oncology, Rotterdam
  - Leyenburg Ziekenhuis; Haematology, The Hague
- New Zealand (3):
  - Auckland city hospital; Auckland Regional Cancer Centre and Blood Service, Auckland
  - Christchurch Hospital; Canterbury Health Laboratories, Christchurch
  - Wellington Hospital; Regional Oncology Unit, Wellington
- Norway (2):
  - Haukeland Universitetshospital; Medicine Dept, Bergen
  - Rikshospitalet Uni Hospital, Oslo
- Poland (6):
  - Medical University School; Dept. of Haematology, Lodz
  - Katedra i Klinika Hematoonkologii i Transplantacji Szpiku; Uniwersytetu Medycznego w Lublinie, Lublin
  - Akademii Medycznej W; Klinika Hematologii, Poznan
  - Klin. Chorob Wewnetrznych I Hemat. Z Osrodkiem Transplant. Szpiku, Warsaw
  - Instytut Hematologii I Transfuzjologii; Klinika Chorob Wewnetrznych I Hematologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny; Haematology Dept., Warsaw
- Romania (4):
  - Fundeni Clinical Inst. ; Hematology Dept, Bucharest
  - Spitalul Clinic Coltea; Clinica de Hematologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu-Mures; compartiment Hematologie, Târgu Mureş
  - Spitalul Clinic municipal de Urgenta Timisoara; Clinica de Hematologie, Timișoara
- Russia (10):
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - Haematology Research Center; Haematology, Moscow
  - City Clinical Botkin's Hospital; City Hematological Center, Moscow
  - Medical Radiological Research Centre Rams; Dept. of Radiotherapy & Chemotherapy of Hemoblastosis, Obninsk
  - Research Inst. Hematology /Blood Transfusion ; Hemablastosis, Supression Hemopoesis & B M Transplant, Saint Petersburg
  - Regional Clinical Hospital; Hematology Dept. #2 For B M Transplantation & High Dose Chemo., Saint Petersburg
  - Pavlov State Medical Uni ; Bone Marrow Transplantation Clinic, Saint Petersburg
  - S.-Peterburg Pavlov State Medical University ; Haematology, Saint Petersburg
  - State Medical Inst. Municipal Hospital #31; Oncology & Hematology Dept. With the Usechemo. in Adult, Saint Petersburg
  - Regional Clinical Hospital N.A. Kalinin; Hematology Dept, Samara
- Spain (5):
  - Hospital Universitario de la Princesa; Servicio de Hematologia, Madrid
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Clinico Universitario de Salamanca;Servicio de Hematologia, Salamanca
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Hematologia, Zaragoza
- Sweden (2):
  - Karolinska Inst. , Huddinge Uni Hospital; Depart. of Hematology, Huddinge
  - Universitetssjukhuset i Linköping, Hematologkliniken, Linköping
- United Kingdom (10):
  - Royal Bournemouth General Hospital; Haematology, Bournemouth
  - Addenbrookes Hospital; Haematology, Cambridge
  - Stobhill Hospital; Dept of Haematology, Glasgow
  - Leeds General Infirmary; Medicine, Leeds
  - Leicester Royal Infirmary; Dept of Haematology, Leicester
  - Royal Liverpool Uni Hospital; Haematology, Liverpool
  - St. Bartholomew'S Hospital; Dept of Medical Oncology, London
  - King'S College Hospital; Haematology, London
  - Royal Marsden Hospital; Academic Dept of Haematology, Sutton
  - Pinderfields General Hospital; Dept of Haematology, Wakefield

REFERENCES:
- [Derived] Weisser M, Yeh RF, Duchateau-Nguyen G, Palermo G, Nguyen TQ, Shi X, Stinson SY, Yu N, Dufour A, Robak T, Salogub GN, Dmoszynska A, Solal-Celigny P, Warzocha K, Loscertales J, Catalano J, Larratt L, Rossiev VA, Bence-Bruckler I, Geisler CH, Montillo M, Fischer K, Fink AM, Hallek M, Bloehdorn J, Busch R, Benner A, Dohner H, Valente N, Wenger MK, Stilgenbauer S, Dornan D. PTK2 expression and immunochemotherapy outcome in chronic lymphocytic leukemia. Blood. 2014 Jul 17;124(3):420-5. doi: 10.1182/blood-2013-12-538975. Epub 2014 Jun 10. PMID 24916506
- [Derived] Dufour A, Palermo G, Zellmeier E, Mellert G, Duchateau-Nguyen G, Schneider S, Benthaus T, Kakadia PM, Spiekermann K, Hiddemann W, Braess J, Truong S, Patten N, Wu L, Lohmann S, Dornan D, GuhaThakurta D, Yeh RF, Salogub G, Solal-Celigny P, Dmoszynska A, Robak T, Montillo M, Catalano J, Geisler CH, Weisser M, Bohlander SK. Inactivation of TP53 correlates with disease progression and low miR-34a expression in previously treated chronic lymphocytic leukemia patients. Blood. 2013 May 2;121(18):3650-7. doi: 10.1182/blood-2012-10-458695. Epub 2013 Mar 22. PMID 23525797

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine+Cyclophosphamide (FC): Fludarabine+cyclophosphamide (FC) intravenously for a total of 6 treatment cycles at intervals of 28 days. Fludarabine: 25 mg/m² IV on Days 1, 2, 3 for 6 cycles. Cyclophosphamide: 250 mg/m² IV on Days 1, 2, 3 for 6 cycles.
- Fludarabine+Cyclophosphamide+Rituximab (FCR): Rituximab and FC intravenously for a total of 6 treatment cycles at intervals of 28 days. Cycle 1: rituximab 375 mg/m² IV on Day 1; fludarabine 25 mg/m² IV on Days 2, 3, 4; cyclophosphamide 250 mg/m² IV on Days 2, 3, 4. Cycles 2-6: rituximab 500 mg/m² IV on Day 1; fludarabine 25 mg/m² IV on Days 1, 2, 3; cyclophosphamide 250 mg/m² IV on Days 1, 2, 3.
Period: Overall Study
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Started | 276 | 276
Safety Population; Received Study Drug | 272 | 274
Completed | 167 (Completed 6 Cycles of Treatment) | 181 (Completed 6 Cycles of Treatment)
Not Completed | 109 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR) | Total
Number analyzed (Participants) | 276 | 276 | 552
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (9.11) | 62.1 (9.17) | 61.7 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 89 | 184
  Male | 181 | 187 | 368

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by the Independent Review Committee (IRC)
Description: Progression-free survival as assessed by the IRC was defined as the time between randomization and the date of first documented disease progression, relapse after response, or death from any cause, whichever came first. Patients without a PFS event were censored at their last tumor assessment date.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: Intent-to-treat (ITT) population was comprised of all patients randomized in the study, irrespective of whether they received treatment or not.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
Days | 660 [556 to 735] | 813 [670 to 947]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); The null hypothesis was that there was no difference between the 2 treatment groups. The alternative hypothesis was that progression-free survival was longer in the fludarabine+cyclophosphamide+rituximab (FCR) group; Test type: Superiority or Other; p = 0.0218, Log Rank; non-stratified; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.60 to 0.96] — The hazard ratio was estimated using Cox regression. The hazard ratio is relative to the fludarabine+cyclophosphamide(FC) group

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was determined from the date of randomization to the date of death irrespective of cause. Patients who had not died at the time of the final analysis (clinical data cut-off) were censored at the date of the last contact.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
Days | 1580 [1408 to NA] — The upper limit could not be estimated due to too low number of events at time of analysis. | NA [1552 to NA] — Median survival time could not be estimated due to too low number of events at time of analysis.
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.2874, Log Rank; non-stratified

3. Secondary Outcome: Number of Participants With Overall Survival (OS) Events
Description: Overall survival was determined from the date of randomization to the date of death (OS event) irrespective of cause. Patients who had not died at the time of the final analysis (clinical data cut-off) were censored at the date of the last contact.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
participants
  Patients with event | 68 | 62
  Patients without events | 208 | 214

4. Secondary Outcome: Event-free Survival (EFS)
Description: Event free survival was measured from the day of randomization to the date of first documented PD, relapse after response, start of a new treatment or death from any cause. Patients without an EFS event were censored at their last tumor assessment date.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
Days | 586 [545 to 731] | 874 [756 to 1187]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0002, Log Rank; non-stratified

5. Secondary Outcome: Number of Participants With Event-free Survival (EFS) Events
Description: Event free survival was measured from the day of randomization to the date of first documented Progressive Disease (PD), relapse after response, start of a new treatment or death from any cause (EFS events). Patients without an EFS event were censored at their last tumor assessment date.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
participants
  Patients with event | 162 | 134
  Patients without events | 114 | 142

6. Primary Outcome: Number of Participants With Progression-free Survival (PFS) Events Assessed by the Independent Review Committee (IRC)
Description: Progression-free survival as assessed by the IRC was defined as the time between randomization and the date of first documented disease progression, relapse after response, or death from any cause (PFS events), whichever came first. Patients without a PFS event were censored at their last tumor assessment date.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
participants
  Patients with event | 148 | 137
  Patients without events | 128 | 139

7. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease free survival was defined for all patients with a best overall response (BOR) of Complete Response (CR) and measured the time from first documented CR in a sequence of consecutive CRs until documented disease progression, relapse or death from any cause. Patients without a DFS event at the time of the analysis (clinical data cut-off) were censored at their last tumor assessment date.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: Intent-to-treat (ITT) population for patients with a Best Overall Response of Complete Response.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 36 | 67
Days | 1285 [791 to NA] — The upper limit could not be estimated due to too low number of events at time of analysis. | 1204 [938 to NA] — The upper limit could not be estimated due to too low number of events at time of analysis.
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.8842, Log Rank; non-stratified

8. Secondary Outcome: Number of Participants With Disease-free Survival (DFS) Events
Description: Disease free survival was defined for all patients with a best overall response (BOR) of Complete Response (CR) and measured the time from first documented CR in a sequence of consecutive CRs until documented disease progression, relapse or death from any cause (DFS events). Patients without a DFS event at the time of the analysis (clinical data cut-off) were censored at their last tumor assessment date.
Time Frame: Mean observation time at time of analysis was approximately 26 months
Population: Intent-to-treat (ITT) population with a Best Overall Response of Complete Response.
Measure: Number; unit: participants
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 36 | 67
participants
  Patients with event | 10 | 19
  Patients without event | 26 | 48

9. Primary Outcome: Final Analysis: Time to Progression-Free Survival Event
Description: Time to progression-free survival (PFS) event was defined as the time between randomization and the date of first documented PFS event: disease progression, relapse or death by any cause, whichever came first.
Time Frame: Median observation time was approximately 5 years
Population: Participants from the Intent-to-treat population, all randomized participants, who experienced a PFS event. Participants who did not have a PFS event at the time of the final analysis were censored at the date of the last contact.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 217 | 205
Days | 683.0 [554 to 797] | 969.0 [809 to 1195]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.54 to 0.80]

10. Secondary Outcome: Final Analysis: Time to Overall Survival Event
Description: Overall survival (OS) was determined from the date of randomization to the date of death (OS event) irrespective of cause.
Time Frame: Median observation time was approximately 5 years
Population: The analysis included only those participants from the Intent-to-treat population,all randomized participants, who died. Participants who had not died at the time of the final analysis were censored at the date of the last contact.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 138 | 144
Days | 2056.0 [1883 to 2344] | 2167.0 [1898 to 2438]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.5976, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.74 to 1.19]

11. Secondary Outcome: Final Analysis: Time to Event-Free Survival Event
Description: Event free survival (EFS) was defined as the time from the day of randomization to the date of first EFS event: documented disease progression, relapse after response, start of a new treatment or death from any cause.
Time Frame: Median observation time was approximately 5 years
Population: Participants from the Intent-to-treat population, all randomized participants, who had an EFS event. Participants who did not have an ESF event at the time of the final analysis were censored at the date of the last contact.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 218 | 207
Days | 630.0 [548 to 747] | 932.0 [777 to 1187]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.54 to 0.79]

12. Secondary Outcome: Final Analysis: Percentage of Participants With Complete Response
Description: Complete response was defined as the disappearance of all signs of cancer in response to treatment.
Time Frame: Median observation time was approximately 5 years
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 276 | 276
Percentage of participants | 13.4 | 25.0
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0005, Chi-squared; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.39 to 3.35]

13. Secondary Outcome: Final Analysis: Time to Disease-Free Survival Event
Description: Time to disease-free survival (DFS) event was defined as the time from first documented response until the first documented DFS event: disease progression, relapse or death from any cause.
Time Frame: Median observation time was approximately 5 years
Population: Participants from the Intent-to-treat population, all randomized participants, with complete response. .
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 37 | 69
Days | 1285.0 [996 to 1541] | 1803.0 [938 to 2071]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.3085, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.46 to 1.28]

14. Secondary Outcome: Final Analysis: Duration of Response
Description: Duration of response was defined as the time between the date of the earliest qualifying response and the date of disease progression or death due to any cause.
Time Frame: Median observation time was approximately 5 years
Population: Participants from the Intent-to-treat population, all randomized participants, with complete or partial response.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 160 | 194
Days | 869.0 [801 to 1107] | 1333.0 [1025 to 1632]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0007, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.51 to 0.84]

15. Secondary Outcome: Final Analysis: Time to New Chronic Lymphocytic Leukemia (CLL) Treatment
Description: Time to new CCL treatment was defined as the time from randomization to the first day of new treatment for CCL or death.
Time Frame: Median observation time was approximately 5 years
Population: Participants from the Intent-to-treat population,all randomized participants, who started a new treatment for CLL or died.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 186 | 173
Days | 1085.0 [997 to 1290] | 1625.0 [1350 to 1805]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.55 to 0.84]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from study start to 28 days after treatment completion (Median observation time= 26 months). Serious Adverse Events were collected 1 year after treatment completion (Median observation time= 37 months).
Description: The safety analysis population included all patients who received at least one dose of trial treatment and had at least one safety follow-up, whether withdrawn prematurely or not. 272 patients received FC only and 274 patients received FCR.
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Serious Adverse Events (participants affected / at risk) | 132/272 | 138/274
Other Adverse Events (participants affected / at risk) | 232/272 | 251/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine+Cyclophosphamide (FC) (N=272) | Fludarabine+Cyclophosphamide+Rituximab (FCR) (N=274)
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Sinusitis (Infections and infestations) | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 11 | 3
Anaemia Haemolytic Autoimmune (Blood and lymphatic system disorders) | 5 | 2
Angina Pectoris (Cardiac disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Aplasia Pure Red Cell (Blood and lymphatic system disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Aspergillosis (Infections and infestations) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Autoimmune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bicytopenia (Blood and lymphatic system disorders) | 2 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 1
Brain Abscess (Infections and infestations) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 6
Bronchitis Viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Chest Wall Abscess (Infections and infestations) | 0 | 1
Chills (General disorders) | 1 | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Coronary Artery Insufficiency (Cardiac disorders) | 1 | 0
Cytomegalovirus Gastrointestinal Infection (Infections and infestations) | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 0
Endocarditis Bacterial (Infections and infestations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Evans Syndrome (Blood and lymphatic system disorders) | 1 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 2 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 21 | 29
Fungal Sepsis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 2
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 5
Herpes Zoster (Infections and infestations) | 3 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection (Infections and infestations) | 3 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Klebsiella Sepsis (Infections and infestations) | 1 | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Listeria Sepsis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung Infection (Infections and infestations) | 1 | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malaise (General disorders) | 1 | 0
Mesenteric Artery Embolism (Gastrointestinal disorders) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycobacterium Avium Complex Infection (Infections and infestations) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Myocardial Infarction (Cardiac disorders) | 2 | 2
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 8
Neutropenic Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 4 | 2
Oral Herpes (Infections and infestations) | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 5 | 5
Parainfluenzae Virus Infection (Infections and infestations) | 1 | 0
Paraneoplastic Pemphigus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Performance Status Decreased (General disorders) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumocystis Jiroveci Infection (Infections and infestations) | 1 | 0
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 18 | 15
Pneumonia Herpes Viral (Infections and infestations) | 0 | 1
Pneumonia Primary Atypical (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pseudomonal Sepsis (Infections and infestations) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 9 | 14
Rectal Abscess (Infections and infestations) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 3 | 4
Septic Shock (Infections and infestations) | 2 | 5
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Supraventricular Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 2
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2
Varicella (Infections and infestations) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
West Nile Viral Infection (Infections and infestations) | 0 | 1
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 0
Capsular Warning Syndrome (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebral Thrombosis (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Nervous System Disorder (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal Failure (Renal and urinary disorders) | 1 | 1
Calculus Ureteric (Renal and urinary disorders) | 1 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Aortic Aneurysm (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Femoral Artery Occlusion (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Peripheral Embolism (Vascular disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Open Wound (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 0
Zygomycosis (Infections and infestations) | 1 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neurological Decompensation (Nervous system disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mycobacterial Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine+Cyclophosphamide (FC) (N=272) | Fludarabine+Cyclophosphamide+Rituximab (FCR) (N=274)
Neutropenia (Blood and lymphatic system disorders) | 110 | 120
Anaemia (Blood and lymphatic system disorders) | 47 | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 33 | 36
Granulocytopenia (Blood and lymphatic system disorders) | 12 | 18
Febrile Neutropenia (Blood and lymphatic system disorders) | 14 | 16
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 23
Bronchitis (Infections and infestations) | 15 | 13
Nasopharyngitis (Infections and infestations) | 15 | 12
Pyrexia (General disorders) | 36 | 60
Fatigue (General disorders) | 45 | 45
Chills (General disorders) | 5 | 41
Asthenia (General disorders) | 30 | 28
Nausea (Gastrointestinal disorders) | 96 | 110
Vomiting (Gastrointestinal disorders) | 50 | 57
Constipation (Gastrointestinal disorders) | 30 | 40
Diarrhoea (Gastrointestinal disorders) | 32 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 34
Headache (Nervous system disorders) | 29 | 25
Hypotension (Vascular disorders) | 2 | 20
Rash (Skin and subcutaneous tissue disorders) | 19 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 20
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 16 | 15
Decreased appetite (Metabolism and nutrition disorders) | 11 | 20
Oedema peripheral (General disorders) | 11 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.